CLINICAL TRIAL: NCT02769962
Title: A Phase I/II Trial of EP0057, a Nanoparticle Camptothecin With Olaparib in Patients With Relapsed/Refractory Small Cell Lung, Bladder and Prostate Cancers
Brief Title: Trial of EP0057, a Nanoparticle Camptothecin With Olaparib in People With Relapsed/Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anish Thomas, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160107; 16-C-0107
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Carcinoma; Urothelial Cancer; Lung Neoplasms; Small Cell Lung Cancer; Prostate Cancer
Keywords: PARP Inhibitor; Topoisomerase I (Top1); Camptothecins; Nanoparticle Drug Conjugate; Solid Tumors
MeSH Terms: conditions — Carcinoma, Transitional Cell; Lung Neoplasms; Small Cell Lung Carcinoma; Prostatic Neoplasms | interventions — IT-101; olaparib; Tomography, X-Ray Computed; Electrocardiography; Echocardiography; Caves; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I - EP0057 (formerly CRLX101) + Olaparib (Experimental): EP0057 + olaparib
  Interventions: Drug: EP0057; Drug: olaparib; Diagnostic Test: CT scan; Diagnostic Test: CT chest, abdomen, and pelvis; Diagnostic Test: Bone scan; Diagnostic Test: ECG; Diagnostic Test: Echocardiogram; Procedure: Biopsy
- 2/Phase II - EP0057 + Olaparib at Maximum Tolerated Dose/Recommended Phase 2 Dose (MTD/RP2D) (Experimental): EP0057 (formerly CRLX101) + olaparib at maximum tolerated dose/recommended phase 2 dose (MTD/RP2D)
  Interventions: Drug: EP0057; Drug: olaparib; Diagnostic Test: CT scan; Diagnostic Test: CT chest, abdomen, and pelvis; Diagnostic Test: Bone scan; Diagnostic Test: ECG; Diagnostic Test: Echocardiogram; Procedure: Biopsy

INTERVENTIONS:
Drug: EP0057 — EP0057 (formerly CRLX101) intravenous (IV) every (Q) 2weeks Day 1 and Day 15, administered in 28-day cycles, until disease progression or development of intolerable side effects.
  Plus olaparib (by mouth (PO) days 3-13* and days 17-26*) administered in 28-day cycles, until disease progression or development of intolerable side effects. Phase (P)1: Dose Escalation P2: recommended phase 2 dose (RP2D).
  (* On days 13 and 26, only one dose of olaparib will be administered in the morning)
  Other Names: CRLX101
Drug: olaparib — Olaparib (by mouth (PO) days 3-13* and days 17-26* administered in 28-day cycles, until disease progression or development of intolerable side effects Plus EP0057 (formerly CRLX101) (intravenous (IV) every (Q) 2 weeks, Day 1 and Day 15) administered in 28-day cycles, until disease progression or development of intolerable side effects. Phase (P)1: Dose Escalation P2: recommended phase 2 dose (RP2D).
  (* On days 13 and 26, only one dose of olaparib will be administered in the morning).
  Other Names: Lynparza
Diagnostic Test: CT scan — Screening and baseline.
  Other Names: Computed tomography scan
Diagnostic Test: CT chest, abdomen, and pelvis — Metastatic castration-resistant prostate cancer (mCRPC) participants only at screening, baseline, cycle 2 Day 1, and end of treatment/disease progression.
Diagnostic Test: Bone scan — Metastatic castration-resistant prostate cancer (mCRPC) participants only at screening, baseline, cycle 2 Day 1, and end of treatment/disease progression.
  Other Names: Bone scintigraphy
Diagnostic Test: ECG — Screening, baseline, Day 1, Day 15 and cycle 2, Day 1.
  Other Names: Electrocardiogram
Diagnostic Test: Echocardiogram — At screening.
  Other Names: Echo
Procedure: Biopsy — Baseline Day 4 and end of treatment/disease progression.

SUMMARY:
Background: EP0057 (formerly CRLX101) consists of a sugar molecule cyclodextrin linked to a chemotherapy drug called camptothecin. The combined molecule or "nanoparticle drug conjugate" travels through the blood. Once inside cancer cells, the chemotherapy drug is released from the molecule. Olaparib is a drug that may stop cancer cells from repairing the deoxyribonucleic acid (DNA) damage caused by chemotherapy. Researchers want to see how safe it is to give EP0057 and olaparib together and to see how well the combination treats a specific type of lung cancer called small cell lung cancer (SCLC).

Objectives:

To test the safety and maximum dose of EP0057 and olaparib together. To test how well they treat small cell lung cancer.

Eligibility:

Adults 18 and older with small cell lung cancer.

Design:

Participants will be screened with standard cancer care tests.

Participants will get the 2 study drugs in 28-day cycles. EP0057 will be given every 2 weeks, through a small plastic tube in an arm vein. Olaparib will be taken by mouth twice a day most days. Participants will keep a pill diary.

For Cycle 1, participants will have 3 visits. All other cycles will have 2 visits.

At study visits, participants may have:

* Blood and hair samples taken
* History and Physical exam
* Questions about health and side effects
* Pregnancy test
* Optional tumor biopsy where a piece of tumor is removed by needle after numbing the skin.
* Computed tomography (CT) scan
* Injection of EP0057 (twice per cycle)
* Olaparib prescription

Participants will have a follow-up visit 4 weeks after finish taking the drugs. They will have a physical exam and blood tests. They may have a tumor biopsy. The study team will call the patient every 3 months for follow up after completing the study treatment.

DETAILED DESCRIPTION:
Background:

* Small cell lung cancer (SCLC) is an aggressive cancer with a poor prognosis.
* Although highly responsive to chemotherapy initially, SCLC relapses quickly and becomes refractory to treatment within a few months.
* Urothelial Carcinoma (UC) of the Bladder is the fourth most common malignancy in men and the ninth most common in women.
* Prostate cancer is the most common cancer among men in the United States. While prostate cancer is initially responsive to androgen deprivation therapy (ADT), the median duration of sensitivity is 24-36 months. Moreover, patients develop resistance to current treatment options.
* The use of poly adenosine diphosphate ribose polymerase (PARP) inhibitors in combination with chemotherapy builds upon pre-clinical data in lung cancer and other cancers supporting the notion that PARP inhibitors potentiate the effect of deoxyribonucleic acid (DNA) damaging therapies.
* Despite their highly synergistic activity in preclinical models, human studies combining PARP inhibitors and camptothecins have not translated into clinical benefit due to enhanced toxicity with the combination.
* One approach to improve ability to combine camptothecins with agents that sensitize their activity like PARP inhibitors is to use alternative formulations that minimize toxicity to the normal tissues.
* EP0057 (formerly CRLX101) is a nanoparticle drug conjugate composed of 20 (S)-camptothecin (a potent and highly selective topoisomerase I inhibitor) conjugated to a linear, cyclodextrin polyethylene glycol-based polymer.
* Olaparib is a PARP inhibitor indicated as monotherapy in patients with deleterious or suspected deleterious germline breast cancer gene (BRCA) mutated advanced ovarian cancer who have been treated with three or more prior lines of chemotherapy. Olaparib has an established safety profile, and it is under investigation in a number of different cancers.

Objectives:

* Phase I: To determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of EP0057 in combination with olaparib in patients with refractory cancers.
* Phase II: To determine the antitumor activity of olaparib plus EP0057 with respect to progression free survival at 16 weeks in SCLC patients with resistant or sensitive relapse.
* Expansion Cohorts: To determine overall response rate of EP0057 plus olaparib in patients with mCRPC and urothelial carcinoma.

Eligibility:

Phase I

* Adult patients >=18 years of age
* Histologically or cytologically confirmed, advanced solid tumor that is refractory to standard therapy and/or for whom no further standard therapy is available
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2

Phase II

* Adult patients >= 18 years old
* Have a pathologically (histology or cytology) confirmed diagnosis of SCLC
* Disease progression on or after at least one platinum-based standard chemotherapy regimen and/or an immune-checkpoint inhibitor for either limited or extensive stage disease.
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* ECOG performance status of 0, 1 or 2

Phase II Expansion Cohorts

* Have a pathologically (histology or cytology) confirmed diagnosis of urothelial carcinoma or metastatic, progressive, castrate resistant prostate cancer (mCRPC)
* Disease progression on or after at least one platinum-based standard chemotherapy regimen and/or an immune-checkpoint inhibitor (except prostate cohort)
* Have measurable disease per RECIST 1.1 (except prostate cohort)
* Prior treatment with enzalutamide and/or abiraterone (prostate cancer cohort only)
* Patients must have castrate levels of testosterone (<50 ng/dl [1.74 nmol/l]) (Prostate cohort only)

Design:

* Patients meeting eligibility criteria will receive EP0057 (intravenous (IV) every (Q) 2weeks) plus olaparib (by mouth (PO) twice a day (BID), days 3-13 and days 17-26 administered in 28-day cycles, until disease progression or development of intolerable side effects. The maximum tolerated dose (MTD) of the combination will be used in Phase II.
* Patients in Phase II will receive, the recommended phase 2 dose (RP2D) at DL4R EP0057 12 mg/m^2 and olaparib 250 mg twice a day (BID).
* Blood, tumor and hair samples will be collected at multiple time points for pharmacokinetics (PK), pharmacodynamics (PD) analyses. Hair sample collection is optional. Tumor biopsies are optional for SCLC and ulcerative colitis (UC) patients and mandatory for metastatic castration-resistant prostate cancer (mCRPC) patients (only baseline biopsy is mandatory).
* Toxicity will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
* Tumor assessments will be made using computed tomography (CT) scans (chest, abdomen and pelvis) at baseline and after every 2 cycles (3 cycles for metastatic castration-resistant prostate cancer (mCRPC) according to RECIST version 1.1.
* After discontinuation of study treatment, follow-up for survival will be carried out every 3 months.

ELIGIBILITY:
* INCLUSION CRITERIA: - Phase I
* Patients must have histologically or cytologically confirmed advanced solid tumor that is resistant or refractory to standard therapy.
* A minimum of 2 weeks will be required from any prior therapy, including chemotherapy, immunotherapy and/or radiation. In addition, recovery to Grade <= 1 from all reversible toxicities related to prior therapy is required at study entry.
* Patients do not need to have measurable disease to enroll on phase I.
* Age 18 years.
* Eastern cooperative Oncology Group (ECOG) performance status <=2
* Patients with treated brain metastases (surgery, whole or stereotactic brain radiation) are allowed provided the lesions have been stable for at least 2 weeks and the patient is off steroids or is on a stable dose of steroids. Patients with brain metastases should not require use of enzyme-inducing antiepileptic drugs (e.g., carbamazepine, phenytoin, or phenobarbital) within 14 days before first dose and during study. Use of newer antiepileptics that do not produce enzyme induction drug-drug interactions (DDIs) is allowed.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >=3,000/mcL
  * absolute neutrophil count >=1,500/mcL without growth factor support
  * platelets >=100,000/mcL without growth factor support
  * hemoglobin >=9 g/dL, and no blood transfusion within 4 weeks.

OR

* Hemoglobin >10 g/dL, and no blood transfusion within 2 weeks.
* total bilirubin <=1.5 x upper limit of normal (ULN) (unless Gilbert's Disease)
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT)<=2.5 X institutional upper limit of normal (<= 5X ULN if liver mets)
* creatinine <= ULN

OR

* creatinine clearance >= 51 mL/min (calculated using the Cockroft-Gault formula) for patients with creatinine levels above institutional normal.

  -The effects of EP0057 (formerly CRLX101) and olaparib on the developing human fetus are unknown. For this reason and because these agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 120 days (both male and female) following last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Fertile females of childbearing potential are defined as women physically capable of becoming pregnant unless the female patient cannot have children because of surgery or other medical reasons (effective tubal ligation, ovaries or the uterus removed, or are post-menopausal). Post-menopausal is defined as:
* Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments,
* Luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for women under 50,
* radiation-induced oophorectomy with last menses >1 year ago,
* chemotherapy-induced menopause with >1 year interval since last menses,
* or surgical sterilization (bilateral oophorectomy or hysterectomy).

  * Negative urine pregnancy test < =3 days prior to cycle 1 day 1 (C1D1) (women of childbearing potential only)
  * Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

INCLUSION CRITERIA: - Phase II Small Cell Lung Cancer (SCLC)

* Age >=18 years.
* Patients must have histologically or cytologically confirmed diagnosis of SCLC from a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
* Have received and progressed during or after a platinum-based standard chemotherapy regimen and/or an immune-checkpoint inhibitor
* Patients could have received any number of therapies for relapsed or progressive disease, including re-treatment with original frontline regimen. A minimum of 2 weeks will be required from any prior therapy, including chemotherapy, immunotherapy and/or radiation. In addition, recovery to Grade <= 1 from all reversible toxicities related to prior therapy is required at study entry. No previous irradiation to the site of measurable or evaluable disease, unless that site had subsequent evidence of progression.
* Patients must have measurable disease as per Response Evaluation Criteria in Solid Tumors, version (RECIST 1.1).
* Radiographic evidence of disease progression after initial therapy should have been documented.
* Eastern Cooperative Oncology Group (ECOG) performance status <=2.
* Patients with treated brain metastases (surgery, whole or stereotactic brain radiation) are allowed provided the lesions have been stable for at least 2 weeks and the patient is off steroids or is on a stable dose of steroids. Patients with brain metastases should not require use of enzyme-inducing antiepileptic drugs (e.g., carbamazepine, phenytoin, or phenobarbital) within 14 days before first dose and during study. Use of newer antiepileptics that do not produce enzyme induction drug-drug interactions (DDIs) is allowed.
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes >=3,000/mcL
  * absolute neutrophil count >=1,500/mcL without growth factor support
  * platelets >=100,000/mcL without growth factor support
  * hemoglobin >=9 g/dL, and no blood transfusion within 4 weeks.

OR

* hemoglobin >10 g/dL, and no blood transfusion within 2 weeks.
* total bilirubin <=1.5 x upper limit of normal (ULN) (unless Gilbert's Disease)
* AST(SGOT)/ALT(SGPT) <=2.5 X institutional upper limit of normal (<= 5X ULN if liver mets)
* creatinine <= ULN

OR

* creatinine clearance >=51 mL/min (calculated using the Cockroft-Gault formula) for patients with creatinine levels above institutional normal.

  * The effects of EP0057 and olaparib on the developing human fetus are unknown. For this reason and because these agents are known to be teratogenic, women of child-bearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 120 days (both male and female) following last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Fertile females of childbearing potential are defined as women physically capable of becoming pregnant unless the female patient cannot have children because of surgery or other medical reasons (effective tubal ligation, ovaries or the uterus removed, or are post-menopausal). Post-menopausal is defined as:
  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments,
* LH and FSH levels in the post-menopausal range for women under 50,
* radiation-induced oophorectomy with last menses >1 year ago,
* chemotherapy-induced menopause with >1 year interval since last menses,
* or surgical sterilization (bilateral oophorectomy or hysterectomy).

INCLUSION CRITERIA: for Urothelial Carcinoma Expansion Cohort (accrual to the cohort ended with amendment version 08/17/2022)

* Patients must have a histologically confirmed diagnosis of urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis from a CLIA-certified laboratory, with measurable disease by RECIST (version 1.1) including lymphadenopathy and visceral metastatic disease
* Male or female patients >= 18 years of age.
* Patient must have received at least one platinum-based regimen of chemotherapy and/or an immune-checkpoint inhibitor if appropriate with progressive disease.
* Prior antiangiogenic and radiation therapy are permitted (2-week washout from therapy is required).
* Bisphosphonates and denosumab are permitted if on a stable dose for >=4 weeks.
* ECOG 0-2

  * Patients must have normal organ and marrow function as defined below:
  * leukocytes >=3,000/mcL
  * absolute neutrophil count >=1,500/mcL without growth factor support
  * platelets >=100,000/mcL without growth
  * factor support
  * hemoglobin >=9 g/dL, and no blood transfusion within 4 weeks.

OR

* hemoglobin >10 g/dL, and no blood transfusion within 2 weeks.
* total bilirubin<TAB> <=1.5 x ULN (unless Gilbert's Disease)
* AST(SGOT)/ALT(SGPT) <=2.5 X institutional upper limit of normal (<= 5X ULN if liver mets)
* creatinine <= ULN

  -The effects of EP0057 and olaparib on the developing human fetus are unknown. For this reason and because these agents are known to be teratogenic, women of child-bearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 120 days (both male and female) following last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Fertile females of childbearing potential are defined as women physically capable of becoming pregnant unless the female patient cannot have children because of surgery or other medical reasons (effective tubal ligation, ovaries or the uterus removed, or are post-menopausal). Post-menopausal is defined as:
* Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments,
* LH and FSH levels in the post-menopausal range for women under 50,
* radiation-induced oophorectomy with last menses >1 year ago,
* chemotherapy-induced menopause with >1 year interval since last menses,
* or surgical sterilization (bilateral oophorectomy or hysterectomy).

  * Patients must be able to tolerate oral medications and not have gastrointestinal illnesses that would preclude absorption of olaparib.
  * Ability to understand and the willingness to sign a written informed consent document.
  * Willingness to release archival tissue sample for research purposes, if available

INCLUSION CRITERIA for mCRPC Expansion Cohort (accrual to the mCRPC cohort ended with amendment version 7/27/2021)

* Patients must have metastatic, progressive, castrate resistant prostate cancer (mCRPC).
* Documented histopathological confirmation of prostate cancer from a CLIA-certified laboratory.
* All patients must have at least one lesion deemed safe to biopsy and be willing to undergo a mandatory baseline biopsy.
* Patients must have received prior treatment with enzalutamide and/or abiraterone with the exception of patients who were treated with docetaxel and androgen deprivation therapy for metastatic castrate-sensitive prostate cancer and progressed on docetaxel treatment or who progress within one month of the last docetaxel dose.
* Patients must have castrate levels of testosterone (<50 ng/dl [1.74 nmol/l])
* Patients must have undergone bilateral surgical castration or must agree to continue on gonadotropin-releasing hormone (GnRH) agonists/antagonists for the duration of the study.
* ECOG performance status <= 2
* Patients must have adequate bone marrow, hepatic, and renal function with:

  * leukocytes >=3,000/mcL
  * absolute neutrophil count >=1,500/mcL without growth factor support
  * platelets >=100,000/mcL without growth factor support
  * Hemoglobin >=9 g/dL, and no blood transfusion within 4 weeks.

OR

* hemoglobin >10 g/dL, and no blood transfusion within 2 weeks.
* total bilirubin <=1.5 x ULN (<=3 (SqrRoot) ULN for subjects with Gilbert's Disease)
* AST(SGOT)/ALT(SGPT) <=3 X institutional upper limit of normal (<= 5X ULN if liver mets)
* creatinine <= ULN

OR

--creatinine clearance >=51 mL/min (calculated using the Cockroft-Gault formula) for patients with creatinine levels above institutional normal.

* Men must be at least 18 years of age.
* Patient must be capable of understanding and complying with protocol requirements and is willing to give informed consent.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of study participation and for 120 days after last dose of study drug. Sexually active subjects and their female partners must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 3 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must also agree to use both a barrier method and a second method of birth control during the course of the study and for 3 months after the last dose of study drug(s). Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.

Patients who were treated for metastatic castrate-sensitive prostate cancer with docetaxel and androgen deprivation therapy who progress on docetaxel treatment or who progress within one month of the last docetaxel dose are eligible.

EXCLUSION CRITERIA: - Phase I and II SCLC and UC Expansion Cohort (note: accrual to the UC cohort ended with amendment version 08/17/2022)

* Patients who are receiving any other investigational agents.
* Persistent toxicities (>= Common Terminology Criteria for Adverse Events (CTCAE) grade 2) with the exception of alopecia and neuropathy, caused by previous cancer therapy
* Patients who have had prior treatment with olaparib or other camptothecin inhibitors (Ulcerative Colitis (UC) expansion Cohort Only).
* Patients with myelodysplastic syndrome/acute myeloid leukemia or active pneumonitis; or baseline features suggestive of myelodysplastic syndrome or acute myelogenous leukemia on peripheral blood smear or bone marrow biopsy, if clinically indicated.
* Hypersensitivity to study therapies ...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2025-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Schmidt KT, Huitema ADR, Dorlo TPC, Peer CJ, Cordes LM, Sciuto L, Wroblewski S, Pommier Y, Madan RA, Thomas A, Figg WD. Population pharmacokinetic analysis of nanoparticle-bound and free camptothecin after administration of NLG207 in adults with advanced solid tumors. Cancer Chemother Pharmacol. 2020 Oct;86(4):475-486. doi: 10.1007/s00280-020-04134-9. Epub 2020 Sep 8. PMID 32897402
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0107.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth): "Confirmed Solid tumor that is resistant or refractory to standard therapy. Drug: EP0057 12mg/m^2 will be administered as an intravenous (IV) infusion over 60-75 minutes every 2 weeks on Day 1 and Day 15 of each cycle.
  Other Names:
  • CLRX101 Pre-medication drugs include a corticosteroid (dexamethasone 20 mg IV) 30-120 minutes prior to start of EP0057, an antihistamine (diphenhydramine 50 mg by mouth (PO), an H2 antagonist (histamine H2-receptor antagonists) (ranitidine 50 mg IV)
  Drug: Olaparib Phase I: A standard 3+3 design will be used, to determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of EP0057 in combination with Olaparib. Phase II: Maximum tolerated dose (MTD) identified in phase I.
  Olaparib 100mg will be given orally twice a day on days 3-13 and days 17-26 administered in 28-day cycles."
- Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth): "Confirmed solid tumor that is resistant or refractory to standard therapy. Drug: EP0057 12mg/m^2 will be administered as an intravenous (IV) infusion over 60-75 minutes every 2 weeks on Day 1 and Day 15 of each cycle.
  Other Names:
  • CLRX101 Pre-medication drugs include a corticosteroid (dexamethasone 20 mg IV) 30-120 minutes prior to start of EP0057, an antihistamine (diphenhydramine 50 mg by mouth (PO), an H2 antagonist (histamine H2-receptor antagonists) (ranitidine 50 mg IV)
  Drug: Olaparib Phase I: A standard 3+3 design will be used, to determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of EP0057 in combination with Olaparib. Phase II: Maximum tolerated dose (MTD) identified in phase I.
  Olaparib 150mg will be given orally twice a day on days 3-13 and days 17-26 administered in 28-day cycles."
- Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth): "Confirmed solid tumor that is resistant or refractory to standard therapy. Drug: EP0057 12mg/m^2 will be administered as an intravenous (IV) infusion over 60-75 minutes every 2 weeks on Day 1 and Day 15 of each cycle.
  Other Names:
  • CLRX101 Pre-medication drugs include a corticosteroid (dexamethasone 20 mg IV) 30-120 minutes prior to start of EP0057, an antihistamine (diphenhydramine 50 mg by mouth (PO), an H2 antagonist (histamine H2-receptor antagonists) (ranitidine 50 mg IV)
  Drug: Olaparib Phase I: A standard 3+3 design will be used, to determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of EP0057 in combination with Olaparib. Phase II: Maximum tolerated dose (MTD) identified in phase I.
  Olaparib 200mg will be given orally twice a day on days 3-13 and days 17-26 administered in 28-day cycles."
- Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth): "Confirmed solid tumor that is resistant or refractory to standard therapy. Drug: EP0057 12mg/m^2 will be administered as an intravenous (IV) infusion over 60-75 minutes every 2 weeks on Day 1 and Day 15 of each cycle.
  Other Names:
  • CLRX101 Pre-medication drugs include a corticosteroid (dexamethasone 20 mg IV) 30-120 minutes prior to start of EP0057, an antihistamine (diphenhydramine 50 mg by mouth (PO), an H2 antagonist H2 antagonist (histamine H2-receptor antagonists) (ranitidine 50 mg IV)
  Drug: Olaparib Phase I: A standard 3+3 design will be used, to determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of EP0057 in combination with Olaparib. Phase II: Maximum tolerated dose (MTD) identified in phase I.
  Olaparib 300mg will be given orally twice a day on days 3-13 and days 17-26 administered in 28-day cycles."
- Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth): "Confirmed Solid tumor that is resistant or refractory to standard therapy. Drug: EP0057 12mg/m^2 will be administered as an intravenous (IV) infusion over 60-75 minutes every 2 weeks on Day 1 and Day 15 of each cycle.
  Other Names:
  • CLRX101 Pre-medication drugs include a corticosteroid (dexamethasone 20 mg IV) 30-120 minutes prior to start of EP0057, an antihistamine (diphenhydramine 50 mg by mouth (PO), an H2 antagonist (histamine H2-receptor antagonists) (ranitidine 50 mg IV)
  Drug: Olaparib Phase I: A standard 3+3 design will be used, to determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of EP0057 in combination with Olaparib. Phase II: Maximum tolerated dose (MTD) identified in phase I.
  Olaparib 250mg will be given orally twice a day on days 3-13 and days 17-26 administered in 28-day cycles."
- Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth): "Small cell lung cancer (SCLC) patients with resistant or sensitive relapse; EP0057 12mg/m^2 will be administered as an intravenous (IV) infusion over 60-75 minutes every 2 weeks on Day 1 and Day 15 of each cycle.
  Other Names:
  • CLRX101 Pre-medication drugs include a corticosteroid (dexamethasone 20 mg IV) 30-120 minutes prior to start of EP0057, an antihistamine (diphenhydramine 50 mg by mouth (PO), an H2 antagonist (histamine H2-receptor antagonists) (ranitidine 50 mg IV)
  Drug: Olaparib Phase II: Maximum tolerated dose (MTD) identified in phase I. Olaparib 250mg will be given orally twice a day on days 3-13 and days 17-26 administered in 28-day cycles."
- Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth): "Confirmed diagnosis of urothelial. Drug: EP0057 12mg/m^2 will be administered as an intravenous (IV) infusion over 60-75 minutes every 2 weeks on Day 1 and Day 15 of each cycle.
  Other Names:
  • CLRX101 Pre-medication drugs include a corticosteroid (dexamethasone 20 mg IV) 30-120 minutes prior to start of EP0057, an antihistamine (diphenhydramine 50 mg by mouth (PO), an H2 antagonist H2 antagonist (histamine H2-receptor antagonists) (ranitidine 50 mg IV)
  Drug: Olaparib Phase I: A standard 3+3 design will be used, to determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of EP0057 in combination with Olaparib. Phase II: Maximum tolerated dose (MTD) identified in phase I.
  Olaparib 250mg will be given orally twice a day on days 3-13 and days 17-26 administered in 28-day cycles."
- Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg: "Confirmed diagnosis of metastatic, progressive, castrate resistant prostate cancer (mCRPC). Drug: EP0057 12mg/m^2 will be administered as an intravenous (IV) infusion over 60-75 minutes every 2 weeks on Day 1 and Day 15 of each cycle.
  Other Names:
  • CLRX101 Pre-medication drugs include a corticosteroid (dexamethasone 20 mg IV) 30-120 minutes prior to start of EP0057, an antihistamine (diphenhydramine 50 mg by mouth (PO), an H2 antagonist H2 antagonist (histamine H2-receptor antagonists) (ranitidine 50 mg IV)
  Drug: Olaparib Phase I: A standard 3+3 design will be used, to determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of EP0057 in combination with Olaparib. Phase II: Maximum tolerated dose (MTD) identified in phase I.
  Olaparib 250mg will be given orally twice a day on days 3-13 and days 17-26 administered in 28-day cycles."
Period: Overall Study
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth) | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Started | 3 | 5 | 3 | 6 | 7 | 13 | 4 | 4
Completed | 3 | 5 | 3 | 6 | 7 | 11 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Refused further treatment | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth) | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg | Total
Number analyzed (Participants) | 3 | 5 | 3 | 6 | 7 | 13 | 4 | 4 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 2 | 4 | 5 | 6 | 4 | 1 | 29
  >=65 years | 1 | 0 | 1 | 2 | 2 | 7 | 0 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.33 (13.32) | 54.2 (2.77) | 61.33 (4.51) | 58.5 (7.45) | 62.43 (7.89) | 63.54 (8.44) | 54.25 (7.85) | 71.25 (10.31) | 61.22 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 3 | 3 | 7 | 0 | 0 | 22
  Male | 0 | 1 | 1 | 3 | 4 | 6 | 4 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 3 | 5 | 3 | 6 | 6 | 13 | 3 | 4 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 5
  White | 2 | 4 | 1 | 6 | 4 | 12 | 4 | 4 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 3 | 6 | 7 | 13 | 4 | 4 | 45

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of EP0057 (CLRX101) in Participants With Refractory Cancers.
Description: MTD/RP2D is the dose level at which no more than 1 of up to 6 participants experience dose-limiting toxicity (DLT) during the DLT evaluation period, and the dose below that at which at least 2 (of ≤6) participants have DLT as a result of the drug. DLTs will be defined using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (Version 4). The following toxicities, occurring during cycle 1 of the study combination, will be considered DLTs if deemed drug-related: Grade 4 neutropenia complicated by fever ≥38.5C and/or documented infection; Grade 4 neutropenia that does not resolve within 7 days; Grade 4 thrombocytopenia that does not resolve within 7 days or grade 3-4 thrombocytopenia complicated with hemorrhage. Grade 4 anemia that does not resolve within 7 days despite optimal therapy; and inability to begin subsequent treatment course within 28 days of the scheduled date, due to study drug toxicity.
Time Frame: First 28 days
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants with solid tumors who received at least one dose of the study drug will be evaluable.
Arm/Group | All Participants
Number analyzed (Participants) | 24
mg/m^2 | 12

2. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of Olaparib in Participants With Refractory Cancers.
Description: as for outcome 1
Time Frame: First 28 days
Measure: Number; unit: mg
Arm/Group | All Participants
Number analyzed (Participants) | 24
mg | 250

3. Primary Outcome: Number of Dose Limiting Toxicities (DLTs) During the First Cycle
Description: DLTs will be defined using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (Version 4). The following toxicities, occurring during cycle 1 of the study combination, will be considered DLTs if deemed drug-related: Grade 4 neutropenia complicated by fever ≥38.5C and/or documented infection; Grade 4 neutropenia that does not resolve within 7 days; Grade 4 thrombocytopenia that does not resolve within 7 days or grade 3-4 thrombocytopenia complicated with hemorrhage. Grade 4 anemia that does not resolve within 7 days despite optimal therapy; and inability to begin subsequent treatment course within 28 days of the scheduled date, due to study drug toxicity, and any Grade 3-4 non-hematologic toxicity except fatigue/asthenia <2 weeks in duration).
Time Frame: First 28 days
Population: Only 23/45 participants were analyzed because DLTs are only completed during phase I. There were only 23 participants in phase I.
Measure: Number; unit: toxicities
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth)
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 7
toxicities | 0 | 0 | 0 | 2 | 1

4. Primary Outcome: Expansion: Progression Free Survival (PFS) Rate in the Combination of Olaparib Plus EP0057 (CLRX101) at 16 Weeks in Small Cell Lung Cancer (SCLC) Participants
Description: Determine if slightly more than 50% of participants may be identified as being without progression by 16 weeks. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 16 weeks
Population: 10/13 participants with small cell lung cancer were analyzed because PFS was only calculated for evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth)
Number analyzed (Participants) | 10
Participants | 2

5. Primary Outcome: Expansion: Overall Response Rate (Complete Response (CR) + Partial Response (PR) of EP0057 (CLRX101) Plus Olaparib in Participants With Urothelial Carcinoma
Description: Overall response rate is the best response recorded from the start of the treatment until disease progression/recurrence. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 8 weeks
Population: 3/4 participants with urothelial carcinoma were analyzed because only 3 of the 4 participants were evaluable; to analyze a response you can only use evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth)
Number analyzed (Participants) | 3
Participants | 1

6. Primary Outcome: Expansion: Overall Response Rate (Complete Response (CR) + Partial Response (PR) of EP0057 (CLRX101) Plus Olaparib in Participants With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Description: Determine if slightly more than 50% of participants may be identified as being without progression by 12 weeks. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 12 weeks
Population: 3/4 participants with metastatic castration-resistant prostate cancer were analyzed because only 3 of the 4 participants were evaluable; to analyze a response you can only use evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Number analyzed (Participants) | 3
Participants | 1

7. Secondary Outcome: Occurrences of Toxicities Including Toxicity Type and Severity (Grades 1, 2, and 3) With Probable Association to Study Regimen in Participants on Expansion Cohorts
Description: Occurrence is captured by subjective and objective data via participant assessment ad self-report. Toxicities including toxicity type and severity (Grades 1, 2, 3, and/or 4) with probable association to study regimen in participants on Expansion cohorts was measured by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening.
Time Frame: Start of treatment through 30 days post last dose, an average of 8.26 months.
Measure: Number; unit: toxicities
Arm/Group | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Number analyzed (Participants) | 13 | 4 | 4
toxicities
  Grade 1 Abdominal pain | 1 | 0 | 0
  Grade 1 Alopecia | 1 | 0 | 1
  Grade 1 Anemia | 1 | 0 | 2
  Grade 1 Anorexia | 1 | 1 | 2
  Grade 1 Constipation | 2 | 0 | 2
  Grade 1 Creatinine increased | 0 | 3 | 2
  Grade 1 Cystitis noninfective | 1 | 0 | 0
  Grade 1 Diarrhea | 3 | 1 | 4
  Grade 1 Dysgeusia | 2 | 0 | 0
  Grade 1 Fatigue | 3 | 0 | 0
  Grade 1 Fever | 0 | 1 | 0
  Grade 1 Gastroesophageal reflux disease | 1 | 0 | 0
  Grade 1 Headache | 0 | 0 | 1
  Grade 1 Hematuria | 1 | 0 | 0
  Grade 1 Hypokalemia | 0 | 1 | 0
  Grade 1 Hyponatremia | 0 | 0 | 1
  Grade 1 Mucositis oral | 0 | 1 | 1
  Grade 1 Myalgia | 0 | 1 | 0
  Grade 1 Nail discoloration | 0 | 0 | 1
  Grade 1 Nausea | 5 | 2 | 2
  Grade 1 Neutrophil count decreased | 1 | 0 | 1
  Grade 1 Platelet count decreased | 3 | 0 | 0
  Grade 1 Stomach pain | 0 | 0 | 1
  Grade 1 Urinary frequency | 0 | 0 | 1
  Grade 1 Urinary tract pain | 0 | 0 | 1
  Grade 1 Vomiting | 4 | 0 | 0
  Grade 1 White blood cell decreased | 5 | 0 | 0
  Grade 2 Abdominal pain | 0 | 1 | 0
  Grade 2 Alopecia | 2 | 0 | 1
  Grade 2 Anemia | 11 | 0 | 1
  Grade 2 Anorexia | 0 | 1 | 0
  Grade 2 Constipation | 1 | 0 | 1
  Grade 2 Creatinine increased | 0 | 4 | 0
  Grade 2 Cystitis noninfective | 1 | 0 | 0
  Grade 2 Diarrhea | 2 | 0 | 0
  Grade 2 Fatigue | 3 | 1 | 3
  Grade 2 Gastroesophageal reflux disease | 1 | 0 | 0
  Grade 2 Infections and infestations - Other specify, oral candidiasis | 0 | 0 | 1
  Grade 2 Lymphocyte count decreased | 9 | 0 | 0
  Grade 2 Mobitz (type) II atrioventricular block | 0 | 0 | 1
  Grade 2 Nausea | 1 | 0 | 1
  Grade 2 Neutrophil count decreased | 4 | 1 | 2
  Grade 2 Platelet count decreased | 1 | 1 | 0
  Grade 2 Proteinuria | 1 | 1 | 0
  Grade 2 Pruritus | 0 | 1 | 0
  Grade 2 Urinary retention | 0 | 0 | 0
  Grade 2 Urinary tract infection | 0 | 0 | 0
  Grade 2 White blood cell decreased | 4 | 1 | 1
  Grade 3 Anemia | 6 | 4 | 1
  Grade 3 Anorexia | 0 | 2 | 0
  Grade 3 Fatigue | 0 | 1 | 1
  Grade 3 Lymphocyte count decreased | 7 | 1 | 0
  Grade 3 Mobitz (type) II atrioventricular block | 0 | 0 | 1
  Grade 3 Platelet count decreased | 1 | 1 | 0
  Grade 3 Thromboembolic event | 0 | 1 | 0
  Grade 3 Urinary tract infection | 0 | 1 | 0
  Grade 3 White blood cell count decreased | 0 | 1 | 1

8. Secondary Outcome: Progression-free Survival (PFS) on Expansion Cohorts
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Every 3 months post-treatment, up until date of death from any cause or an average of 9.57 months.
Population: 16/21 participants in the expansion cohort were analyzed because this was the number of evaluable participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Number analyzed (Participants) | 10 | 3 | 3
Months | 1.97 [0.95 to 10.41] | 1.90 [1.37 to 7.32] | 8.67 [1.8 to 19.48]

9. Secondary Outcome: Progression-free Survival (PFS) of the Combination
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Duration of time from start of treatment to time of progression or death, whichever occurs first, up to 2.5 years
Population: 18/24 participants with solid tumors were analyzed because these were the evaluable participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 5
Months | 4.71 [2.63 to 7.18] | 8.37 [3.16 to 30.36] | 8.37 [3.16 to 30.36] | 4.154 [2.24 to 6.59] | 13.18 [3.82 to 22.35]

10. Secondary Outcome: Overall Survival (OS) of the Combination
Description: OS is defined as the date of on-study to the date of death from any cause or last follow up.
Time Frame: Date of on-study to the date of death from any cause or last follow up, up to 2.5 years
Population: 34/45 participants were analyzed because these were the evaluable participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth) | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 5 | 10 | 3 | 3
Months | 2.07 [1.91 to 2.83] | 2.30 [1.87 to 5.53] | 2.57 [2.34 to 6.09] | 1.54 [0.98 to 3.26] | 9.72 [2.04 to 13.87] | 4.15 [1.54 to 73.16] | 5.88 [4.59 to 25.45] | 14.02 [12.91 to 19.48]

11. Secondary Outcome: Prostate-specific Antigen (PSA) on Metastatic Castration-Resistant Prostate Cancer (mCRPC) Expansion Cohort Reported at Time of Documented Partial Response (PR) With an 80% Confidence Interval
Description: PSA levels in blood, date of cycle 1, Day 1 (C1D1) - Best response date. PSA levels were measured by the Enzyme-Linked Immunosorbent Assay (ELISA). Normal PSA level is ≤6.5 ng/mL for age 70-79 and an elevated level is not interpreted good or bad; a very high number is a strong indicator of prostate cancer; since this is a cohort of prostate cancer an elevated number is expected. Partial Response was assessed by the Response Evaluation Criteria in Solid Tumors in Solid Tumors (RECIST) guideline (version 1.1) and Prostate Cancer Clinical Trials Working Group criteria (PCWG2). Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 40.71 weeks from start of treatment to best response date
Population: 1/4 participants were analyzed because they were not evaluable.
Measure: Number (80% Confidence Interval); unit: ng/mL
Arm/Group | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Number analyzed (Participants) | 1
ng/mL
  C1D1 PSA | 75.35 [NA to NA] — An 80% confidence interval cannot be calculated from just one observation because there is no way to estimate variability or the spread of the data.
  Best Response date PSA | 32.14 [NA to NA] — An 80% confidence interval cannot be calculated from just one observation because there is no way to estimate variability or the spread of the data.

12. Secondary Outcome: Prostate-specific Antigen (PSA) on Metastatic Castration-Resistant Prostate Cancer (mCRPC) Expansion Cohort Reported at Time of Documented Partial Response (PR) an 95% Confidence Interval
Description: PSA levels in blood were measured by the Enzyme-Linked Immunosorbent Assay (ELISA). Normal PSA level is ≤6.5 ng/mL for age 70-79 and an elevated level is not interpreted good or bad; a very high number is a strong indicator of prostate cancer; since this is a cohort of prostate cancer an elevated number is expected; it is noted that this number is decreased from the start of therapy. Partial Response was assessed by the Response Evaluation Criteria in Solid Tumors in Solid Tumors (RECIST) guideline (version 1.1) and Prostate Cancer Clinical Trials Working Group criteria (PCWG2). Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 40.71 weeks from start of treatment to best response date.
Measure: Number (95% Confidence Interval); unit: ng/mL
Arm/Group | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Number analyzed (Participants) | 1
ng/mL
  C1D1 PSA | 75.35 [NA to NA] — A 95% confidence interval and median cannot be calculated from just one observation because there is no way to estimate variability or the spread of the data.
  Best Response date PSA | 32.14 [NA to NA] — A 95% confidence interval and median cannot be calculated from just one observation because there is no way to estimate variability or the spread of the data.

13. Secondary Outcome: Duration of Response (DOR) of the Combination
Description: DOR is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. OS is determined from the start of treatment until death. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: At baseline and after every 2 cycles up until the date of first documented progression or an average of average 11.09 months.
Population: 5/45 participants were analyzed because only 5/45 participants were evaluable.
Measure: Median (Full Range); unit: Months
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth) | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Months |  |  |  |  | 7.95 [7.85 to 8.04] | NA [lower limit 5.05] — Median and upper end of confidence of confidence interval cannot be estimated for one participant. | NA [lower limit 2.75] — Median and upper end of confidence of confidence interval cannot be estimated for one participant. | NA [lower limit 10.11] — Median and upper end of confidence of confidence interval cannot be estimated for one participant.

14. Secondary Outcome: Occurrences of Toxicities Including Toxicity Type and Severity (Grades 1, 2, 3, 4 and/or 5) With Probable Association to Study Regimen in Participants on Solid Tumor Cohorts
Description: Occurrence is captured by subjective and objective data via participant assessment and self-report. Toxicities including toxicity type and severity (Grades 1, 2, 3, and/or 4) with probable association to study regimen in participants on Expansion cohorts was measured by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to adverse event (AE).
Time Frame: Start of treatment through 30 days post last dose, up to 3.99 months
Measure: Number; unit: occurrences of toxicities
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth)
Number analyzed (Participants) | 3 | 5 | 3 | 6 | 7
occurrences of toxicities
  Grade 1 Abdominal pain | 0 | 0 | 0 | 0 | 1
  Grade 1 Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 2
  Grade 1 Alkaline phosphatase increased | 0 | 0 | 0 | 0 | 2
  Grade 1 Alopecia | 0 | 0 | 0 | 0 | 4
  Grade 1 Anemia | 1 | 3 | 5 | 1 | 12
  Grade 1 Anorexia | 0 | 0 | 0 | 2 | 3
  Grade 1 Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 1
  Grade 1 Bloating | 0 | 1 | 0 | 1 | 0
  Grade 1 Constipation | 0 | 0 | 0 | 0 | 3
  Grade 1 Cough | 0 | 0 | 0 | 0 | 1
  Grade 1 Creatinine increased | 1 | 1 | 0 | 5 | 3
  Grade 1 Cystitis noninfective | 0 | 0 | 0 | 0 | 1
  Grade 1 Diarrhea | 0 | 0 | 0 | 0 | 3
  Grade 1 Dizziness | 0 | 0 | 0 | 0 | 2
  Grade 1 Dysgeusia | 0 | 0 | 0 | 0 | 3
  Grade 1 Dyspepsia | 1 | 1 | 0 | 1 | 0
  Grade 1 Dysphagia | 0 | 0 | 0 | 0 | 1
  Grade 1 Fatigue | 0 | 1 | 1 | 1 | 3
  Grade 1 GGT increased | 0 | 0 | 0 | 0 | 1
  Grade 1 Headache | 0 | 0 | 0 | 0 | 1
  Grade 1 Hypokalemia | 0 | 1 | 0 | 2 | 54
  Grade 1 Hypomagnesemia | 0 | 1 | 0 | 0 | 1
  Grade 1 Lymphocyte count decreased | 3 | 10 | 4 | 11 | 11
  Grade 1 Nausea | 0 | 0 | 2 | 2 | 6
  Grade 1 Neutrophil count decreased | 0 | 1 | 5 | 2 | 2
  Grade 1 Platelet count decreased | 2 | 2 | 3 | 10 | 13
  Grade 1 Sore throat | 0 | 0 | 0 | 0 | 1
  Grade 1 Urinary retention | 0 | 0 | 0 | 1 | 0
  Grade 1 Urinary tract pain | 0 | 0 | 0 | 1 | 1
  Grade 1 Vaginal pain | 0 | 0 | 0 | 0 | 1
  Grade 1 Vomiting | 0 | 1 | 1 | 0 | 3
  Grade 1 White blood cell decreased | 1 | 3 | 10 | 3 | 12
  Grade 2 Abdominal pain | 0 | 0 | 0 | 0 | 1
  Grade 2 Alopecia | 0 | 0 | 0 | 0 | 0
  Grade 2 Anemia | 3 | 8 | 7 | 6 | 20
  Grade 2 Anorexia | 0 | 0 | 0 | 0 | 3
  Grade 2 Constipation | 0 | 0 | 0 | 0 | 1
  Grade 2 Cough | 0 | 0 | 0 | 0 | 0
  Grade 2 Creatinine increased | 0 | 0 | 0 | 0 | 0
  Grade 2 Diarrhea | 0 | 0 | 0 | 0 | 1
  Grade 2 Dyspepsia | 0 | 0 | 0 | 0 | 1
  Grade 2 Fatigue | 1 | 0 | 0 | 2 | 0
  Grade 2 Gastroesophageal reflux disease | 0 | 0 | 0 | 0 | 1
  Grade 2 Hypophosphatemia | 0 | 0 | 0 | 2 | 1
  Grade 2 Infusion related reaction | 3 | 0 | 0 | 0 | 0
  Grade 2 Lung infection | 0 | 0 | 0 | 0 | 1
  Grade 2 Lymphocyte count decreased | 1 | 6 | 3 | 12 | 18
  Grade 2 Nausea | 0 | 0 | 0 | 0 | 3
  Grade 2 Neutrophil count decreased | 1 | 2 | 4 | 7 | 5
  Grade 2 Pain in extremity | 0 | 0 | 0 | 0 | 1
  Grade 2 Platelet count decreased | 2 | 1 | 3 | 3 | 2
  Grade 2 Sinus tachycardia | 0 | 0 | 0 | 1 | 0
  Grade 2 Upper respiratory infection | 0 | 0 | 0 | 0 | 1
  Grade 2 Urinary tract infection | 0 | 0 | 0 | 0 | 1
  Grade 2 Vaginal pain | 0 | 0 | 0 | 0 | 1
  Grade 2 Vomiting | 0 | 0 | 0 | 0 | 0
  Grade 2 White blood cell decreased | 2 | 2 | 6 | 8 | 9
  Grade 3 Anemia | 0 | 1 | 5 | 4 | 9
  Grade 3 Febrile neutropenia | 0 | 0 | 0 | 0 | 1
  Grade 3 Lymphocyte count decreased | 0 | 0 | 3 | 3 | 13
  Grade 3 Neutrophil count decreased | 0 | 1 | 1 | 6 | 3
  Grade 3 Platelet count decreased | 1 | 0 | 1 | 2 | 3
  Grade 3 Vomiting | 0 | 0 | 0 | 0 | 1
  Grade 3 Weight loss | 0 | 0 | 0 | 0 | 1
  Grade 3 White cell count decreased | 1 | 1 | 3 | 3 | 4
  Grade 4 Lymphocyte count decreased | 1 | 0 | 2 | 0 | 0
  Grade 4 Neutrophil count decreased | 0 | 0 | 0 | 4 | 5
  Grade 4 Platelet count decreased | 1 | 0 | 1 | 1 | 1
  Grade 4 White blood cell count decreased | 0 | 0 | 2 | 2 | 3
  Grade 5 Any toxicity | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Maximum Observed Plasma Concentration of EP0057 (Both the Total Drug and Released Camptothecin) and Olaparib
Description: Blood samples for pharmacokinetic (PK) analysis were collected at pre-dose, mid-infusion (30 minutes), end of infusion (EOI), and 1, 2, 12, 24, and 48 hours (hr) post-EOI. Samples were drawn into sodium heparin tubes, processed to plasma, and stored at -80°C. On Cycle 6 Day 1 (C6D1), additional samples were collected to evaluate EP0057 (CLRX101) accumulation and potential drug interactions. Total plasma concentrations of released camptothecin (CPT) were measured after acidification with 0.1 normality (N) hydrochloric acid (HCl) to stabilize the lactone form, followed by dilution and Ultra-Performance Liquid Chromatography-Tandem Mass Spectrometry, (UPLC-MS/MS) analysis. Noncompartmental analysis was used to calculate PK parameters. Concentrations below lower limit of quantification (LLOQ) was excluded. Maximum serum concentration (CMAX) values were recorded as observed.
Time Frame: Cycle 1 (pre-dose, mid-infusion (30 minutes), end of infusion (EOI), and 1, 2, 12, 24, and 48 hours (hr) post-EOI); and Cycle 6 Day 1.
Population: 24/45 participants were analyzed because pharmacokinetics for phase II was not collected. These were not collected for Ph II as they were in the study calendar of the protocol for Phase I. This outcome was only calculated for phase I solid tumors. 2/3 participants were analyzed in solid tumor dose level 1 because one participant was omitted due to incomplete serial PK collection.
Measure: Mean (Standard Deviation); unit: Ng/mL
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth)
Number analyzed (Participants) | 2 | 5 | 3 | 6 | 7
Ng/mL
  EP0057 Total Drug | 6191.2 (354.01) | 5641.1 (682.36) | 5307.0 (475.81) | 4998.4 (538.03) | 5844.9 (797.76)
  EP0057 Released Camptothecin | 403.61 (63.307) | 355.14 (116.03) | 332.24 (76.841) | 168.03 (82.751) | 205.10 (59.736)
  Olaparib | 2843.0 (947.62) | 1773.9 (1548.0) | 4729.8 (2375.2) | 5238.6 (4132.4) | 5445.7 (4865.5)

16. Secondary Outcome: Pharmacodynamic (PD) Activity of EP0057 in Surrogate Tissue Specimens
Description: Drug concentrations in tissue specimens.
Time Frame: Baseline, Cycle 1, then every 2 cycles, and at progression
Reporting Status: Not Posted, anticipated posting 2027-07

17. Secondary Outcome: Pharmacodynamic (PD) Activity of EP0057 in Tumor Biopsy Specimens
Description: Drug concentrations in tumor specimens.
Time Frame: Baseline, Cycle 1, then every 2 cycles, and at progression
Population: Data was collected for 4 participants but not analyzed. We will never submit results because PD evaluation cannot be performed on baseline biopsies. Pharmacodynamic studies aim to assess the biological effects of a drug on its target or pathway within the tissue after administration. Baseline biopsies, collected prior to any treatment, reflect the untreated state of the tissue and therefore do not provide information on drug-induced changes or target modulation.
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth) | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse Events was monitored/assessed from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent (s) was/were administered, an average of 6.08 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth) | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
Number analyzed (Participants) | 3 | 5 | 3 | 6 | 7 | 13 | 4 | 4
Participants | 3 | 5 | 3 | 6 | 7 | 13 | 4 | 4

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed an average of 9.57 months. Adverse Events was monitored/assessed from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent (s) was/were administered, an average of 6.08 months.
Description: Adverse Events will be recorded from the first study intervention, Study Day 1, through 30 days after the last study drug administration. Adverse events that are serious need to be recorded through 30 days after the last study drug administration. Beyond 30 days after the last study drug administration and through the end of study participation, only adverse events which are serious and related to the study intervention need to be recorded.
Arm/Group | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth) | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg
All-Cause Mortality (participants affected / at risk) | 3/3 | 5/5 | 3/3 | 6/6 | 7/7 | 11/13 | 4/4 | 4/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/5 | 1/3 | 6/6 | 6/7 | 6/13 | 3/4 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 3/3 | 6/6 | 7/7 | 13/13 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) (N=3) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) (N=5) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) (N=3) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) (N=6) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth) (N=7) | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) (N=13) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) (N=4) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify: Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify: C diff (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — - Other, specify: Malignant pleural mesothelioma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — - Other, specify: Newly detected right frontal parietal brain mass
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — - Other, specify: Progressive Disease
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — - Other, specify: Progressive disease
Nervous system disorders - Other, specify: Left lower extremity numbness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify: Word finding difficulty (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Redness of mediport area (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Tumor Dose Level 1: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 100mg (by Mouth) (N=3) | Solid Tumor Dose Level 2: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 150mg (by Mouth) (N=5) | Solid Tumor Dose Level 3: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 200mg (by Mouth) (N=3) | Solid Tumor Dose Level 4: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 300mg (by Mouth) (N=6) | Solid Tumor Dose Level 4R: EP0057 (CLRX101) 12mg/m^2 (Intravenous); Olaparib 250mg (by Mouth) (N=7) | Small Cell Lung Cancer Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) (N=13) | Urothelial Carcinoma Dose Level 4R:EP0057(CLRX101) 12mg/m^2(Intravenous); Olaparib 250mg(by Mouth) (N=4) | Metastatic Castration-Resistant Prostate Cancer Dose Level 4R: EP0057 12mg/m^2; Olaparib 250mg (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (6) | 3 (4) | 2 (3) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 5 (8) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (3) | 1 (1) | 2 (2) | 4 (7) | 7 (18) | 2 (2) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (3) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 3 (15) | 2 (17) | 5 (11) | 6 (43) | 6 (19) | 1 (2) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (9) | 3 (4) | 2 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 5 (9) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (4) | 2 (5) | 2 (2) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (2) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (7) | 7 (8) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 1 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 2 (3) | 1 (1) | 3 (8) | 2 (5) | 0 (0) | 3 (6) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 5 (9) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (4) | 1 (1) | 2 (2)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 10 (10) | 2 (2) | 2 (4)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Black stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify: Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify: Night sweats (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — - Other, specify: Intrahepatic and extrahepatic biliary ductal dilation secondary to external compression
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 3 (6) | 2 (3) | 5 (16) | 7 (17) | 2 (2) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 3 (5) | 1 (2) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 1 (1) | 3 (7) | 4 (13) | 5 (7) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (7) | 1 (3) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: C diff (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (7) | 5 (19) | 3 (12) | 6 (26) | 5 (42) | 5 (17) | 1 (2) | 0 (0)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Cramping in L hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 4 (9) | 5 (7) | 2 (4) | 3 (3)
Nervous system disorders - Other, specify: Muscle jerks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (4) | 3 (10) | 5 (18) | 4 (14) | 3 (5) | 1 (1) | 1 (3)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (6) | 1 (3) | 2 (8) | 5 (17) | 5 (19) | 3 (8) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Urine output decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — - Other, specify: Around the ankles- redness with no pain or itching. Possibly r/t walking in thick grass
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — - Other, specify: Lump on chest Left lower back(hip) and right ankle
Skin and subcutaneous tissue disorders - Other, specify: Rash: b/l LLE- no itching, not painful. (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Rash: rt shoulder, dry skin. (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 4 (5) | 3 (4) | 1 (2) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (4) | 3 (6) | 3 (21) | 5 (16) | 5 (28) | 3 (11) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT02769962/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT02769962/ICF_001.pdf